CLINICAL TRIAL: NCT02001428
Title: Intermittent Screening and Treatment for the Control of Malaria in the First Year of Life in Papua, Indonesia: A Cluster Randomized Controlled Trial
Brief Title: Malaria in Early Life Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Timika Research Facility, Indonesia (Unknown); Eijkman Institute for Molecular Biology (Other); Menzies School of Health Research (Other)
Responsible Party: Principal Investigator, Dr. Jeanne Rini Poespoprodjo, Maternal and Child Health Consultant, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WT099875_Malaria in Early Life
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Plasmodium Falciparum Malaria; Plasmodium Vivax Malaria
Keywords: malaria; vivax; falciparum; infants
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent Screening and Treatment (Experimental): Infants enrolled at Village health posts will be randomly allocated to receive intermittent screening and treatment (IST) on every scheduled immunization visit at 2, 3, 4 and 9 months of age. Infants in this group will be screened for malaria by Rapid Diagnostic Test (RDT), and if positive, treated with dihydroartemisinin-piperaquine (DHP). Infants will also receive follow up home visits at 6 and 12 months.
  Interventions: Drug: dihydroartemisinin-piperaquine
- Passive Case Detection (No Intervention): Infants in the control arm will only be checked for malaria if they have fever, or history of fever in the 24 hours prior to the scheduled immunization visit at 2,3,4 and 9 months of age, or at a follow up home visit at 6 and 12 months. Infants with malaria will be treated with DHP once daily for 3 days according to local treatment guidelines.

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — Participating infants with uncomplicated malaria will be treated with a three day course (1 dose/day) of DHP (containing 40 mg dihydroartemisinin and 320 mg piperaquine) administered as a total dose over three days of 6mg/kg of dihydroartemisinin and 57 mg/kg of piperaquine.
  Other Names: DHP
  Arms: Intermittent Screening and Treatment

SUMMARY:
The purpose of this study is to assess the effectiveness of different malaria control strategies in the first year of life.

The effectiveness of delivering an intermittent screening and treatment programme with dihydroartemisinin-piperaquine (DHP), linked to local immunization programmes, will be compared to the current practice of passive case detection of malaria.

This study has two objectives:

1. To assess the effectiveness of intermittent screening and treatment with dihydroartemisinin-piperaquine (DHP) administered at 2, 3, 4 and 9 months of age compared with the current practice of passive detection and treatment for malaria in an area with high drug resistance levels to both P. falciparum and P. vivax.
2. To evaluate the safety, efficacy and population pharmacokinetics of DHP in children under 1 year of age.

DETAILED DESCRIPTION:
Infant malaria is a major public health issue in Timika, Papua (Indonesia) and the risk starts at birth with the majority of malaria, mostly asymptomatic, in the first 3 days of life. Malaria infection is associated with severe complications, such as severe anaemia and respiratory distress, and can be fatal.

The emergence of multidrug resistant malaria poses a significant health risk to this vulnerable group. In addition, due to non-specific symptoms of malaria found in this age group, the diagnosis is often missed. Early detection and prompt treatment with an effective antimalarial drug is the key to prevent adverse outcomes from malaria in the first year of life.

The first line treatment for uncomplicated malaria in Indonesia is Dihydroartemisinin-piperaquine (DHP), an ACT that has been shown to be highly efficacious in this region, although experience of its use in infants less than one year old is limited.

Although the World Health Organization recommends antimalarial drug efficacy trials in infants, most ACT efficacy studies include children aged one year or older. Drug population pharmacokinetic studies have enrolled younger infants aged 5-6 months old, whereas Intermittent Preventive Treatment in Infants (IPTi) studies usually start with infants as young as 3 months old.

In view of the challenges to identifying an effective malaria treatment for infants in Indonesia, the proposed study has been designed to evaluate the effectiveness of delivering early detection and prompt treatment with DHP at 2, 3, 4 and 9 months of age, linked to local immunization programmes delivered at village health posts (Posyandu), in an area with high drug resistance levels to both P. falciparum and P. vivax. The effectiveness of this approach will be compared to the current practice of passive case detection. We will also define the efficacy and pharmacokinetic profile of DHP in infancy and monitor the safety and toxicity of its use.

The proposed study will enrol 756 infants across 5 health centres in Papua, Indonesia. Infants will be recruited from pregnant mothers who are enrolled as participants of the concurrent STOPMiP trial - a clinical research study which aims to evaluate intermittent screening and treatment (IST) or intermittent preventive therapy (IPT) with DHP in pregnant women in Indonesia.

The trial result will inform policy makers in Indonesia, and internationally, on the effectiveness of different malaria control strategies in the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Mother of participant is enrolled in the STOP MiP trial
* Healthy full term newborn of consenting parent
* Residence in the study area for the duration of the follow up period

Exclusion Criteria:

* Preterm infants (<37 weeks gestation)
* Sick newborns, requiring hospitalization

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 757 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
The incidence of clinical malaria in the first year of life | Total number of new clinical cases per child during the first year of life
  The total number of new clinical malaria cases from birth to one year old will be measured at one year of age.

SECONDARY OUTCOMES:
Proportion of infant with recurrent parasitaemia due to any species at day 42 after treatment with DHP. | Parasitaemia found at day 42 after treatment with DHP
  Malaria parasitaemia is assessed by microscopy and PCR.

OTHER OUTCOMES:
Prevalence of anaemia and malaria at 6 and 12 months of age. | Prevalence will be assessed at 6 and 12 months of age
Population mean pharmacokinetic profile of Piperaquine | the piperaquine level will be assessed at day 0,1,2,7,14,21,28,35 and 42 after treatment with DHP
  Key pharmacokinetic parameters, CL/F (clearance relative to bioavailability), Vss/F (Volume of distribution at steady state relative to bioavailability), t½,z (elimination half life) will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne R Poespoprodjo, MD, MSc, PhD, Principal Investigator — University of Gadjah Madah
Locations (1):
- Timika Research Facility, Timika, Special Region of Papua, Indonesia

REFERENCES:
- [Derived] Poespoprodjo JR, Hafiidhaturrahmah, Sariyanti N, Indrawanti R, McLean ARD, Simpson JA, Kenangalem E, Burdam FH, Noviyanti R, Trianty L, Fadhilah C, Soenarto Y, Price RN. Intermittent screening and treatment for malaria complementary to routine immunisation in the first year of life in Papua, Indonesia: a cluster randomised superiority trial. BMC Med. 2022 Jun 8;20(1):190. doi: 10.1186/s12916-022-02394-1. PMID 35672703
- See also: Registration information for the related STOP MiP clinical trial — http://www.controlled-trials.com/ISRCTN34010937/